CLINICAL TRIAL: NCT01300104
Title: Feasibility Study on a Nordic Lifestyle Intervention Trial Investigating the Effect of Vigorous Activity and Intake of Whole Grain Rye on Cancer Progression, Insulin Sensitivity and Inflammation Among Men With Early Stage Prostate Cancer.
Brief Title: Feasibility Study on a Nordic Lifestyle Intervention Trial Among Men With Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Cancer Society (Other)
Collaborators: Aarhus University Hospital (Other); University of Aarhus (Other); European Commission (Other)
Responsible Party: Principal Investigator, Rikke Dalgaard Hansen, Principal Investigator / Project Manager, Danish Cancer Society
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC Grant agreement 242244; CHANCES (Other Grant/Funding Number: European Commission)
Record Dates: First submitted 2011-02-18; First posted 2011-02-21 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2015-02

CONDITIONS: Prostate Cancer
Keywords: prostate cancer progression; active surveillance; whole grain rye; exercise; insulin sensitivity; quality of life
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity; Insulin Resistance | interventions — Exercise; Health Planning Guidelines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise and whole grain rye (Experimental)
  Interventions: Behavioral: Exercise; Behavioral: Whole grain rye; Behavioral: Recommendations
- No prescriptions (Active Comparator)
  Interventions: Behavioral: Recommendations

INTERVENTIONS:
Behavioral: Exercise — Prescriptions: Vigorous exercise (average 65-70% of maximal oxygen consumption) minimum 3 times 45 minutes per week according to customized endurance training programs.
  Restrictions: None.
  Arms: Exercise and whole grain rye
Behavioral: Whole grain rye — Prescriptions: Minimum 170-180g of whole grain rye intake per day. Restrictions: None.
  Arms: Exercise and whole grain rye
Behavioral: Recommendations — Recommendations on a health-promoting, energy restricted diet according to Danish Nutrition Recommendations and encouraged to walk at least 10,000 steps every day.

SUMMARY:
PURPOSE:

To evaluate the feasibility of a future Nordic intervention trial, including vigorous activity and a high intake of whole grain rye, among prostate cancer patients on active surveillance.

Additionally, to investigate effects of the lifestyle intervention according to cancer progression, the metabolic profile, inflammation and quality of life among prostate cancer patients on active surveillance.

DETAILED DESCRIPTION:
In the present feasibility study it will be established whether it is possible to enroll participants for this particular kind of intervention among this particular patient group, and if compliance with the intervention is possible to gain by the tools planned: individual counselling with a dietician and a physiologist, interviews on diet, exercise tests and diaries on diet, exercise and steps taken.

Furthermore, the investigators will investigate if we are able to detect effects of the lifestyle intervention according to cancer progression, the metabolic profile, inflammation and quality of life among the participants (24 men) within the short intervention period (6 months) for this particular feasibility study.

Biomarkers of effect and compliance are measured in blood, urine and prostate tissue samples. Metabolomics and the following biomarkers are measured in blood and urine samples: Alkyl resorcinols, enterolactone, tnf receptor 2, e-selectin. ICAM1, IL1-alpha, IL6, triglycerides, HDL/LDL, s-insulin, HbA1c, C-peptide, CRP, IGF1, GLP1, cholesterol, cathepsin and glucose.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven prostate cancer within 2 years prior to enrolment
* PSA ≤ 10 ng/ml, Gleason-score ≤ 6, clinical localized prostate cancer ≤ cT2a or PSA ≤ 10 ng/ml, Gleason-score ≤ 7, clinical localized prostate cancer ≤ cT2a.
* Maximum 1/5 tumor positive biopsy rate
* On active surveillance (elected to forgo treatment)
* Level of testosterone normal in sera

Exclusion Criteria:

* Prior history of cancer, except for non-melanoma skin cancer, unless considered cured without signs of treatment failure for at least five years
* Less than 10 years of life expectancy
* Conditions or behaviors likely to affect the capability of participating fully in the intervention
* Moderate to severe co-morbidity (kidney, liver, heart or respiratory problems) or the general physical constitution
* Gluten intolerance
* Inflammatory bowel disease (e.g. Crohn, colitis)
* Physical handicaps

Ages: 55 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of a planned Nordic life style intervention | Five years
  Feasibility of an intervention trial is evaluated among Danish men with early stage prostate cancer. Enrollment of participants, possible for this particular type of trial among the particular patient group? Compliance with intervention, obtainable for intervention participants with the tools planned (counseling sessions, exercise programs, supply of rye products, sphygmographs and pedometers)? Does the design minimize drop out? Is the schedule for monitoring, counseling, testing and collection of biological samples efficient and feasible for the research team and for the participants?

SECONDARY OUTCOMES:
Prostate cancer progression, effect of the life style intervention | One year
  PSA is measured at baseline and 3, 6 and 12 months after baseline among all participants. Prostate biopsies are made at baseline and 6 months after baseline among all participants.
Insulin sensitivity and insulin secretion, effect of the life style intervention | One year
  Oral glucoce tolerance test is made among all participants at baseline, and 3, 6 and 12 months after baseline.
  C peptide levels will be measured in 24h urine samples the following year after the intervention. The urine samples are collected at baseline, and 3, 6 and 12 months after baseline from all participants.
Life quality, effect of the life style intervention | One year
  Life quality is evaluated by questionnaires answered by all participants at baseline, and 6 and 12 months after baseline.
Metabolic profile, effect of the life style intervention | One year
  The following measurements are made at baseline, and 3, 6 and 12 months after baseline among all participants: Bioimpedance, skin fold analysis, waist and hip circumference, weight and height, and blood pressure.
Inflammation, effect of the life style intervention | One year
  CRP is measured among all participants at baseline, and 3, 6 and 12 months after baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Tjønneland, Dr.Med.Sci., Study Director — Danish Cancer Society Research Center; Rikke D Hansen, Dr., Principal Investigator — Danish Cancer Society Research Center; Michael Borre, Prof., Study Director — Aarhus University Hospital Skejby
Locations (4):
- Denmark (4):
  - Aarhus University, Institute of Sport Science, Aarhus
  - Counseling Center, Danish Cancer Society, Aarhus
  - Aarhus University Hospital Skejby, Aarhus
  - Danish Cancer Society, Copenhagen

REFERENCES:
- [Derived] Eriksen AK, Hansen RD, Borre M, Larsen RG, Jensen JM, Overgaard K, Borre M, Kyro C, Landberg R, Olsen A, Tjonneland A. A lifestyle intervention among elderly men on active surveillance for non-aggressive prostate cancer: a randomised feasibility study with whole-grain rye and exercise. Trials. 2017 Jan 13;18(1):20. doi: 10.1186/s13063-016-1734-1. PMID 28086943